CLINICAL TRIAL: NCT00832689
Title: Irinotecan, Gemcitabine, Chemotherapy for Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Seung Woo Park, Professor, Severance hospital
Purpose: Treatment
Other Study IDs: 4-2007-0191
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Biliary Tract Cancer
Keywords: toxicity
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Irinotecan; Gemcitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Irinotecan and Gemcitabine

INTERVENTIONS:
Drug: Irinotecan and Gemcitabine

SUMMARY:
The study hypothesis is that chemotherapy of irinotecan and gemcitabine will improve local control of cancer and prolong survival in patients with inoperable biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed inoperable biliary tract cancer
* Age: 18 ~75 years old
* Performance status: ECOG 0-2
* Hematopoietic:

  * Granulocyte count at least 1,500/mm3
  * Platelet count at least 100,000/mm3
* Hepatic:

  * Bilirubin No greater than 2 fold the upper normal limit
  * AST/ALT : No greater than 3 fold the upper normal limit
* Renal:

  * Creatinine - no greater than 1.5 mg/dL
* Not pregnant
* No other serious medical or psychiatric illness that would preclude giving informed consent or limit
* No prior chemotherapy within 6 months
* No other concurrent anticancer radiotherapy within 6 months

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Youp Park, MD, Study Director — Assistant professor of division of Gastroenterology
Locations (1):
- Severance hospital, Seoul, South Korea